CLINICAL TRIAL: NCT04061785
Title: Impact of Skills Acquired Through Judo Training on Risk Factors for Falling in Elderly Men and Women
Acronym: J4BE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna University (Other)
Collaborators: The Swedish Judo Federation (Unknown); Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Michail Tonkonogi, Professor, Dalarna University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: J4B190723
Record Dates: First submitted 2019-08-14; First posted 2019-08-20 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Aging Problems; Frailty; Fall Injury; Accidental Fall; Fear of Falling
Keywords: Fall prevention; Physical training; judo; exercise; Judo4Balance; Break falls; Preventive Exercise
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants in 12 week Judo Inspired Exercise program (Active Comparator): The subjects will participate in a 12 week judo inspired training program (45 minute sessions once a week) with the specific aim to increase physical qualities related to falls and injuries during falls.
  The subjects will be tested before and after the 12 week period
  Interventions: Other: Judo4Balance - 12 week judo inspired exercise program
- Control Group (No Intervention): The subjects will go about their normal life for 12 weeks without any intervention. The persons will be tested before and after the 12 week period.

INTERVENTIONS:
Other: Judo4Balance - 12 week judo inspired exercise program — 12 weeks x 45 minute judo inspired exercise in lead by instructor in a group setting.
  Arms: Participants in 12 week Judo Inspired Exercise program

SUMMARY:
Falls and injuries from falls are one of the greatest threats to public health. One of the risk factors for accidental falls is a low self-efficacy regarding the perceived capability to perform activities without the risk of falling. Judo is a sport which include "break fall" strategies where falls with correct landing strategies and rolling movements are in focus in order to avoid injuries. The investigators expect that a judo inspired training (Judo4Balance) will strengthen self-efficacy when it comes to the perceived ability to perform daily tasks without the risk of falling and thereby reduce the risk for falling. Judo based training also includes a well rounded training with focus on strength, balance, explosive power, stamina, proprioception and flexibility. These physical qualities are of importance for reducing the risk of falling. Therefore the investigators' hypothesis is that a 12 week long judo inspired training program could be a suitable tool for reducing falls.

The aim of the project is to evaluate and document whether a 12 week standardized judo inspired exercise program including both the training of above mentioned physical qualities as well as "break fall" techniques can influence the risk of falling as well as reduce the negative consequences such as injuries from an accidental fall.

For the evaluation of the 12 week intervention a validated test battery will be used which gives an indication of the risk for falling in the near future. Furthermore, a specifically designed "Falling Competence" Test has been developed by the investigators' M. Tonoknogi and K Strömqvist Bååthe to measure "break fall" technique.

If it can be proven that the intervention group reaches the expected positive results then the control group will be offered the same type of Judo4Balance training after that they have been participating as a randomized control group.

There is evidence that the risk of falling can be reduced by training, nevertheless judo based training has not to the investigator's knowledge been scientifically investigated among the elderly with the aim of reducing the risk of falls. Neither has it been studied if this type of group training is motivational for continuing physical activity after the intervention.

Due to the Covid-19 pandemic and the Swedish Govt. recommendations (in mid March 2020) to avoid group exercises for older adults (to decrease the risk of the spread of Covid-19) the 9 exercise intervention groups where put on hold/paused after 6-9 weeks into the exercise program.

We applied for and received an approval for an addition to the ethical approval (2019-03048), in order to follow up with the study subject after 6-7 months of self-quarantine in the homes with a self rating of: Fall EfficacyScale (FES), EQ3D as well as questionnaire about the subjects perceived physical and mental health. These questionnaires were sent by post.

DETAILED DESCRIPTION:
The aim of this study is to evaluate and document whether a 12 week standardized judo based exercise program which include both the physical as well as "break fall" technique can influence the risk of falling as well as reduce the negative consequences of an accidental fall.

Questions asked:

* Can a 12 week standardized judo based exercise program improve the physical status with regard to risks for falls among elderly ?
* Can a 12 week standardized judo based exercise program improve the balance among elderly.
* Can a 12 week standardized judo based exercise program improve the self-efficacy among elderly so they can perform their daily chores without the fear of falling
* Can a 12 week standardized judo based exercise program increase the level of physical activity among elderly?
* Can a 12 week standardized judo based exercise program decrease the risk of falls among elderly?
* Is there a difference between men and women regarding the effects on fall rate and on physical factors influencing fall injuries after the completed sixteen week standardized judo based training program

The intervention study is conducted in cooperation with the Swedish Judo Federation who has developed as standardized exercise program for the elderly named Judo4Balance. The recommended training is well in accordance with the physical exercises that are intrinsic to a judo practice. Therefore the hypothesis is that a 12 week long judo inspired training program could be a suitable tool for reducing falls and injuries from falls.

For the evaluation of the 12 week intervention a validated test battery which gives an indication of the risk of falling for an individual in the near future will be used. There will also be a specifically designed Falling Competence test to measure the effectiveness of the "break fall" training.

Furthermore a follow up of the participants' physical status and break fall technique as well as their level of physical activity will be conducted with the same set of tests two years after the first intervention.

The persons included in the study will where it is possible be followed up regarding fall incidents for several years.

If it can be proven that the intervention group reaches the expected positive results such as improved physical status, higher self-efficacy with regards to falling and increased technical "break fall" skills then the control group will be offered the same type of Judo4Balance training one or two terms after that they have been participating as a randomized control group.

There is evidence that the risk of falling can be reduced by training, nevertheless judo based training has not to the investigators's knowledge been scientifically investigated among the elderly with the aim of reducing the risk of falls. Neither has it been studied if this type of group training is motivational for continuing physical activity after the intervention.

A randomized control study consisting of an intervention study and a control group that is carried out between 2019 - 2022 at different places throughout Sweden.

Recruitment will be made at local health centers, judo clubs, and through cooperation with clubs and activity centers for retired people.

Older adults interested in the intervention will be informed about the study both in written form and verbally and are signing a consent form. Independent research assistants perform the tests. After the tests are made the participants in the study will be randomized into one of two groups. One group will participate in the standardized judo inspired 12 week practice and one group will not participate. Practical tests and questionnaires are repeated again after the 12 weeks regardless of group affiliation.

The judo based exercise program (Judo4Balance)is divided into three blocks and is lead by experienced and especially trained judo teachers during 12 - 16 weeks (12 -16 sessions)

Block 1) Good technique during break fall training and strength training, accustom the body to regular training, find the right level of training for the group, build up load resistance in muscles, tendons and bones, challenge the balance through new movements that are not used during daily living activities such as getting down and up from the floor, flexibility training för stiff joints such as neck, upper back and shoulders.

Block 2) Improve "break fall" technique and strength exercises, increase the load in the strength exercises, challenge the balance and coordination, increase the range of motion, introduce "power" exercises when the participants master the technique, continue to build up the load resistance in muscles, tendons, and bones.

Block 3) Train the skill of explosive power during strength exercises and break falls. Challenge the balance with increased complexity and difficulty.

Before the intervention and after the 12 week of standardized judo training program and for the control group no specific program given the following tests will be made:

The participants fill in a health declaration and a questionnaire that besides demographic information also includes questions about motivation through two questions regarding readiness for change and self-efficacy regarding performing daily tasks without fear of falling.

Modified Falls-Efficacy Scale - Swedish version (FES(S)) is a validated questionnaire which measures the self confidence in performing an activity without falling on an 11 grade scale, where 0 is not sure at all and 10 is totally confident when performing the activity without falling. The participant rates oneself based on 13 described activities where maximum score is 130 points.

The physical status with relevance to fall risk will be evaluated using the modified Short Physical Performance Battery (SPPB) where each physical function, balance, strength and walking is evaluated on a 4 grade scale. The test has a max points of 12 and has proven to have a good reliability according to test - retest.

The Mini-Balance Evaluation System Test (Mini-BESTest) is used to measure balance. The test includes 14 different tasks on 4 sub-scales. All tasks are graded from 0 to 2 points, with a total maximum score of 28 points. The test has high reported test-retest reliability and inter rater reliability.

Since there are no previously known tests for the evaluation of judo "break fall" techniques for adults or elderly people, two tests have been designed by Professor M. Tonkonogi & Research Assistant K. Strömqvist Bååthe at Dalarna University in cooperation with The Swedish Judo Federation to test the acquired skills for falling backwards as well as falling forwards in a safe setting, with progressive difficulty. The judo fall techniques are graded on a 0-4 scale. Where 0 represents the minimum score and 4 the maximum score. Four judo puzzle mats are needed for the exercises.

Frändin/Grimby Activity Scale will be used to measure the level of physical activity. The scales range from 1 to 6, with 1 representing 'hardly active at all' and 6 representing 'intensive exercise regularly and several times per week.' The scale has been evaluated and shown to have good validity.

European Quality of Life Questionnaire (EQ-5D or EQ3D) will be used to measure quality of life in five dimensions, hygiene, main activities, pain, worry and mood/depression. Furthermore an evaluation of the participant's health status is made on a vertical analogue scale (VAS) graded 0-100. EQ-5D is proven to have a good test-retest reliability and a high validity.

The pattern of movement will be analyzed before, and after the intervention with the help of "surface - electromyograph electrodes placed bilaterally on the participant's back muscles and accelerometer based mobility sensors placed on the perons's wrists, ankles and chest.

Change over time will be calculated with paired non-parametric statistics for nominal and original data. Change over time for interval and quote data is calculated with parametric statistics. Uni-variate data and multivariate data analysis will be used for calculating change and outcome variables between the groups over time A p-Value <0.05 is needed to show a significant difference.

The study had to be temporarily suspended because of the Covid pandemic after 6-9 sessions. However, in the fall of 2021 we were able to restart the training with both the exercise group as well as the control group. Both groups trained for 12 weeks. The test battery was performed both before and after the 12 week intervention.

ELIGIBILITY:
Inclusion Criteria:

* 55 - 110 years of age
* Understanding oral and written communication in Swedish

Exclusion Criteria:

* Cannot sit up without support
* Not being able to hold up neck when laying on the floor or rolling backwards.
* Aortic aneurysm,
* Angina pectoris
* Cataract operation within the last 6 months

Ages: 55 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in "break fall" competence/skills | Before and after 12 weeks
  Two tests by the name "Judo4Balance - Falling Competence Test" - Backward and forward have been developed to test skills for falling backwards as well as falling forwards in a safe setting, with progressive difficulty. The judo "break-fall technique is graded on a 0-4 scale where 0 represents the minimum score and 4 represents the maximum score for each test .
  Minimum Score = 0 = The subject is unable to lay down on the mat and lift the head from the surface and then stand up independently.
  Maximum Score = 4 = the subejct is able to fall backwards or forwards from a standing up position without any dangerous maneuver
  * A dangerous maneuver is an action which could during a fall increase the risk of injury such as: not holding up the head, not lowering the center of gravity, putting out hand or elbow etc. If a dangerous maneuver is spotted the test will be stopped.
Change in Participants' Falls Efficacy after 12 weeks | Before and after 12 weeks of training (+addition after 7 months of self quarantine)
  The change in participants' falls-efficacy will be measured through - Modified Falls-Efficacy Scale - Swedish version (FES(S))A validated questionnaire which measures the self confidence in performing an activity without falling on an 11 grade scale, where 0 is not sure at all and 10 is totally confident when performing the activity without falling.The subject rates oneself based on 13 described activities where maximum score is 130 points.

SECONDARY OUTCOMES:
Change in Physical Function, Balance, Strength and Walking | Before and after 12 weeks
  This outcome will be measured through: Short Physical Performance Battery (SPPB)A test where each physical function, balance, strength and walking is evaluated on a 4 grade scale. The test has a max points of 12 and has proven to have a good test-retest reliability.
Change in Balance | Before and after 12 weeks
  The Mini-Balance Evaluation Test (Mini-BEST)- Is a test used to measure balance. The test includes 14 different tasks on 4 subscales. All tasks are graded from 0 to 2 points, with a total maximum score of 28 points. The test has high reported test-retest reliability and interrater reliability.
Change in level of Physical Activity | Before and after 12 weeks (+addition after 7 months of self quarantine after Covid pandemic)
  Frändin/Grimby Activity Scale will be used to measure the level of physical activity. The scales range from 1 to 6, with 1 representing 'hardly active at all' and 6 representing 'intensive exercise regularly and several times per week.' The scale has been evaluated and shown to have good validity.
Change in Quality of Life | Before and after 12 weeks (+addition after 7 months of self quarantine during Covid pandemic)
  European quality of life questionnaire (EQ-3D) will be used to measure quality of life in five dimensions, hygiene, main activities, pain, worry and mood/depression. Furthermore an evaluation of the persons health status is made on a vertical analogue s (VAS) graded 0-100. EQ-5D is proven to have a good test-retest reliability and a high validity.
Identification of depressive symptoms after quarantine the last 2 weeks | (addition after 7 months of self quarantine)
  WHO 5

OTHER OUTCOMES:
Change in movement patterns when having fear of falling | Before and after 12 weeks
  Optional on some of the subjects.
  The participant's pattern of movement will be analyzed before, and after the intervention with the help of "surface-Electromyography (EMG) electrodes place bilaterally on the back muscles and accelerometer based mobility sensors placed on the participants's wrists, ankles and chest.

CONTACTS AND LOCATIONS:
Overall Officials: Michail Tonkonogi, PhD, Principal Investigator — Dalarna University
Locations (1):
- Dalarna University, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Timsina LR, Willetts JL, Brennan MJ, Marucci-Wellman H, Lombardi DA, Courtney TK, Verma SK. Circumstances of fall-related injuries by age and gender among community-dwelling adults in the United States. PLoS One. 2017 May 4;12(5):e0176561. doi: 10.1371/journal.pone.0176561. eCollection 2017. PMID 28472065
- [Background] Hellström K, Sandström M, Heideken Wågert P, et al. Fall-Related Self-efficacy in Instrumental Activities of Daily Living is Associated with Falls in Older Community-Living People. Phys Occup Ther Geriatr. 2013;31(2):128-139.
- [Background] Franchini, E, Kiss, MA, Sterkowicz S. Physical fitness and anthropometrical differences between elite and non elite judo players. Biol Sport 2005; 22: 315-328, 2005.
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Frändin K, Grimby G. Assessment of physical activity, fitness and performance in 76-year-olds. Scand J Med Sci Sports. 1994; 4(1), 41
- [Background] Hellstrom K, Lindmark B, Wahlberg B, Fugl-Meyer AR. Self-efficacy in relation to impairments and activities of daily living disability in elderly patients with stroke: a prospective investigation. J Rehabil Med. 2003 Sep;35(5):202-7. doi: 10.1080/16501970310000836. PMID 14582550
- [Background] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Derived] Arkkukangas M, Stromqvist Baathe K, Ekholm A, Tonkonogi M. Short Multicomponent Group Exercise Intervention Promotes Long-Term Physical Activity Habits among Community-Dwelling Older Adults during COVID-19 Restrictions: A Cohort Study. Int J Environ Res Public Health. 2022 Nov 17;19(22):15140. doi: 10.3390/ijerph192215140. PMID 36429859
- See also: Description and film from the Swedish Judo4Balance exercise program for elderly — https://judo.se/fallprevention/falltrygghet-for-aldre/